CLINICAL TRIAL: NCT01035138
Title: Open-Label Extension for Alzheimer's Disease Patients Who Complete One of Two Semagacestat Phase 3 Double-Blind Studies (H6L-MC-LFAN or H6L-MC-LFBC)
Brief Title: A Study of Semagacestat for Alzheimer's Patients
Acronym: Identity XT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5930; H6L-MC-LFBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N2-((2S)-2-(3,5-difluorophenyl)-2-hydroxyethanoyl)-N1-((7S)-5-methyl-6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-L-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: semagacestat (Experimental)
  Interventions: Drug: semagacestat

INTERVENTIONS:
Drug: semagacestat — 140mg administered orally, once daily for 24 months; dose reduction to 100mg or 60 mg possible due to intolerability
  Other Names: LY450139

SUMMARY:
The primary objective of the original study was to assess the safety of semagacestat in Alzheimer's disease (AD) patients during 24 months of open-label treatment. Baseline for the efficacy measures is defined as the baseline for feeder studies LFAN (NCT00594568) and LFBC (NCT00762411). For all safety analyses (adverse events), baseline for patients will be week 0 of this study (LFBF).

Preliminary results from LFAN and LFBC showed semagacestat did not slow disease progression and was associated with worsening of clinical measures of cognition and the ability to perform activities of daily living. Study drug was stopped in all studies. Studies LFAN, LFBC and LFBF have been amended to continue collecting safety data, including cognitive scores, for at least seven months. The CT-Registry will reflect results of analyses from the original protocol in addition to those from the amended protocol. Very few participants from LFBC rolled over into LFBF (N = 9). Due to insufficient sample size, the data for LFBC participants who rolled into LFBF were not analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Meets National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable Alzheimer's Disease
* Completed semagacestat study LFAN or study LFBC through 88 weeks
* Must continue to have a reliable caregiver
* Capable of swallowing whole oral medication
* Agrees not to participate in other investigational compounds for the duration of study

Exclusion Criteria:

* Meets LFAN or LFBC study discontinuation criteria at the last visit of the LFAN or LFBC study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (71):
- United States (41):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sun City, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Costa Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lomita, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooksville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deerfield Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa Bay, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyannis, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jenkintown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bennington, Vermont
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geelong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg West, Victoria
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Penticton, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Chile (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antofagasta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdivia
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse, France
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siegen
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashkelon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan, Italy
- Japan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellville, South Africa
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plasencia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- LFAN Placebo/LY140 mg: Participants received placebo orally once daily for 76 weeks during study LFAN. At the end of 76 weeks, participants received LY450319 titrated up to 140 milligram (mg) orally once daily. Participants continued 140 mg LY450319 (LY 140 mg) orally once daily up to 24 months during this extension study (LFBF)
- LFAN LY 100 mg/ LY 140 mg: Participants received 100 mg LY450319 (LY 100 mg) orally once daily during study LFAN, and 140 mg LY450319 orally once daily up to 24 months during this extension study (LFBF)
- LFAN LY 140 mg/LY 140 mg: Participants received 140 mg LY450319 orally once daily during study LFAN, and 140 mg LY450319 orally once daily up to 24 months during this extension study (LFBF)
Period: Overall Study
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Started | 73 | 60 | 47
Completed | 0 | 0 | 0
Not Completed | 73 | 60 | 47
Not completed — Adverse Event | 4 | 0 | 2
Not completed — Caregiver Decision | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Sponsor Decision | 66 | 60 | 42
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- LFAN Placebo/LY140 mg: Participants received placebo orally once daily for 76 weeks during study LFAN. At the end of 76 weeks, participants received LY450319 titrated up to 140 mg orally once daily. Participants continued 140 mg LY450319 (LY 140 mg) orally once daily up to 24 months during this extension study (LFBF)
- LFAN LY 100 mg/ LY 140 mg: Participants received 100 mg LY450319 orally once daily during study LFAN, and 140 mg LY450319 orally once daily up to 24 months during extension study
- LFAN LY 140 mg/LY 140 mg: Participants received 140 mg LY450319 orally once daily during study LFAN, and 140 mg LY450319 orally once daily up to 24 months during extension study
- Total: Total of all reporting groups
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg | Total
Number analyzed (Participants) | 73 | 60 | 47 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.3) | 73.5 (8.7) | 74.1 (9.5) | 73.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 33 | 21 | 93
  Male | 34 | 27 | 26 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  White | 61 | 58 | 42 | 161
  Black or African American | 2 | 0 | 0 | 2
  Asian | 8 | 2 | 4 | 14
  Multi-racial | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 29 | 107
  Finland | 3 | 0 | 0 | 3
  Spain | 2 | 2 | 2 | 6
  Chile | 1 | 2 | 0 | 3
  Israel | 2 | 1 | 2 | 5
  Italy | 1 | 0 | 0 | 1
  France | 2 | 0 | 0 | 2
  Canada | 4 | 5 | 3 | 12
  Poland | 0 | 0 | 2 | 2
  Australia | 3 | 3 | 0 | 6
  South Africa | 1 | 0 | 0 | 1
  Germany | 8 | 5 | 5 | 18
  Japan | 6 | 2 | 3 | 11
  Sweden | 0 | 2 | 1 | 3
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog11) [Mean (Standard Deviation); unit: units on a scale] — The cognitive subscale of the ADAS (ADAS-Cog11) was used as a primary efficacy measure and consisted of 11 items assessing areas of function most typically impaired in AD: orientation, verbal memory, language, and praxis. The scale ranged from 0-70, with higher scores indicating greater disease severity.
  units on a scale | 21.0 (8.5) | 21.1 (8.5) | 21.5 (9.3) | 21.1 (8.7)
Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) [Mean (Standard Deviation); unit: units on a scale] — The ADCS-ADL was a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. It measures both basic and instrumental activities of daily living. The total ADCS-ADL score ranged from 0-78, with lower scores indicating greater disease severity.
  units on a scale | 63.7 (11.4) | 65.5 (9.0) | 62.2 (12.2) | 63.9 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog11) at Week 16 After Cessation of Study Drug
Description: The cognitive subscale of the ADAS (ADAS-Cog11) consists of 11 items assessing areas of function most typically impaired in Alzheimer's Disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity.
Time Frame: Baseline (LFAN randomization), 16 weeks (LFBF) after cessation of study drug
Population: Participants who completed Study LFAN, took at least one dose of study drug in extension study and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 41 | 40 | 26
units on a scale | 6.4 (11.53) | 12.5 (12.82) | 10.5 (13.62)

2. Primary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) at Week 16 After Cessation of Study Drug
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. It measures both basic and instrumental activities of daily living. The total score ranges from 0 to 78, with lower scores indicating greater disease severity.
Time Frame: Baseline (LFAN randomization), 16 weeks (LFBF) after cessation of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 36 | 33 | 21
units on a scale | -4.5 (7.73) | -10.6 (15.15) | -5.1 (11.28)

3. Secondary Outcome: Percent Change From Baseline in Amyloid Beta (Aβ) 1-42 Plasma Concentration at Week 12
Description: Concentration of amino acid peptide known as Aβ 1-42 in plasma. Least Square (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (LFAN Randomization ), 6 hours pose-dose at Week 12 (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 11 | 18 | 7
percentage of change | -5.84 (16.03) | -6.09 (9.01) | 14.27 (17.37)

4. Secondary Outcome: Change From Baseline in Hippocampal Volume Using Volumetric Magnetic Resonance Imaging (vMRI) at Week 12
Description: The vMRI assessment of right hippocampal and left hippocampal volume is reported. Least Square (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cubic millimeter (mm³)
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 9 | 7 | 3
cubic millimeter (mm³)
  Left hippocampal volume | -115.39 (83.61) | -279.29 (77.55) | 22.49 (107.49)
  Right hippocampal volume | -141.79 (81.00) | -187.16 (65.53) | -3.86 (99.85)

5. Secondary Outcome: Change From Baseline in Amyloid Imaging Positron Emission Tomography (AV-45-PET) at Week 12
Description: A radioactive tracer for PET that is a ligand for amyloid called [18F]-AV-45. This permits the visualization of amyloid in the brains of Alzheimer's participants. The outcome reported is the composite summary of the standard uptake value ratio for the cerebellar gray matter. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator. Due to insufficient sample size, this analysis was not done.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: Due to insufficient sample size, this analysis was not done.
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog11) at Week 12
Description: The cognitive subscale of the ADAS (ADAS-Cog11) consists of 11 items assessing areas of function most typically impaired in Alzheimer's Disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. Least Square (LS) Mean value was controlled for baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 65 | 53 | 43
units on a scale | 9.3 (1.52) | 8.06 (1.67) | 11.56 (1.79)

7. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog12) at Week 12
Description: ADAS-Cog12 is the ADAS-Cog11 augmented with the delayed free recall measure, resulting in a total score ranging from 0 to 80. Higher scores indicate greater disease severity. Least Square (LS) Mean value was controlled for baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 65 | 53 | 43
units on a scale | 10.35 (1.60) | 9.09 (1.75) | 12.66 (1.88)

8. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog14) at Week 12
Description: The ADAS-Cog14 is the ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity. Least Square (LS) Mean value was controlled for the baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 65 | 52 | 43
units on a scale | 11.31 (1.78) | 10.02 (1.99) | 14.50 (2.10)

9. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) at Week 12
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. It measures both basic and instrumental activities of daily living. The total score ranges from 0 to 78, with lower scores indicating greater disease severity. Least Square (LS) Mean value was controlled for baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 60 | 50 | 36
units on a scale | -12.34 (2.11) | -8.22 (2.36) | -8.74 (2.67)

10. Secondary Outcome: Mean Concentration of LY450139
Time Frame: 3 months (pre-dose, 2, 4, and 6 hours after dosing )(LFBF)
Population: Participants who completed Study LFAN, took study drug in extension study and had pharmacokinetics measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- LY 140 mg: Participants received 140 mg LY450319 orally once daily up to 24 months during extension study (LFBF)
Arm/Group | LY 140 mg
Number analyzed (Participants) | 46
nanogram/milliliter (ng/mL)
  Pre-dose (n=7) | 1.81 (124)
  2 hours after dosing (n=46) | 1160 (66.9)
  4 hours after dosing (n=44) | 679 (41.9)
  6 hours after dosing (n=41) | 341 (52.6)

11. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog12) at Week 16 After Cessation of Study Drug
Description: ADAS-Cog12 is the ADAS-Cog11 augmented with the delayed free recall measure, resulting in a total score ranging from 0 to 80. Higher scores indicate greater disease severity.
Time Frame: Baseline (LFAN Randomization), 16 weeks (LFBF) after cessation of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 41 | 40 | 26
units on a scale | 6.7 (12.05) | 12.6 (13.11) | 11.2 (14.97)

12. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog14) at Week 16 After Cessation of Study Drug
Description: The ADAS-Cog14 is the ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity.
Time Frame: Baseline (LFAN Randomization), 16 weeks (LFBF) after cessation of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 41 | 40 | 26
units on a scale | 7.7 (13.21) | 14.1 (14.66) | 13.3 (16.93)

13. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Scale (Sum of Boxes) (CDR-SB) at Week 24
Description: The CDR-SB is a semi-structured interview of participants and their caregivers. The participant's cognitive status is rated in 6 domains of functioning, including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. A severity score is assigned for each of the 6 domains with total score ranging from 0 to 18. Higher scores indicate greater disease severity. Least Square (LS) Mean value was controlled for baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 24 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 63 | 52 | 39
units on a scale | 4.18 (0.53) | 2.99 (0.58) | 3.39 (0.65)

14. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) at Week 24
Description: The MMSE is a brief screening instrument used to assess cognitive function in elderly participants. It assesses orientation, memory, attention, and ability to name objects, follow verbal and written commands, write a sentence, and copy figures. The total score ranges from 0 to 30, with a lower score indicating greater disease severity. Least Square (LS) Mean value was controlled for baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 24 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 62 | 51 | 41
units on a scale | -4.67 (0.78) | -4.15 (0.85) | -4.84 (0.91)

15. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) at Week 24
Description: The NPI is a tool for assessing psychopathology in patients with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the patient's behavior. The score ranges from 12 to 144, with higher scores indicating greater disease severity. Least Square (LS) Mean value was controlled for the baseline value, age, investigator, concomitant standard of care medication.
Time Frame: Baseline (LFAN Randomization), 24 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 18 | 23 | 9
units on a scale | 1.87 (4.68) | 1.94 (3.62) | 3.62 (6.43)

16. Secondary Outcome: Change From Baseline in EuroQol-5D (EQ-5D) at Week 24
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression; each has 3 severity levels (no, some, severe problems) coded to a 1-digit number (1-3). Digits are combined into 5-digit number describing health state. Numbers 1-3 are not added for total score. Visual Analog Scale (VAS) assesses caregiver's impression of participant's overall health state; VAS scores range=0-100, with lower scores indicating greater disease severity. LS Mean value was controlled for baseline value, age, investigator, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (LFAN Randomization), 24 weeks (LFBF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 62 | 54 | 42
units on a scale | 0.76 (3.19) | -2.23 (3.38) | -14.44 (3.67)

17. Secondary Outcome: Change From Baseline in Resource Utilization in Dementia-Lite Questionnaire (RUD-Lite) at Week 12
Description: RUD-Lite assesses the healthcare resource utilization of participants and their caregivers to determine the level of formal and informal care attributable to Alzheimer's Disease (AD). Information on both caregivers (caregiving time, work status) and participants (accommodation and healthcare resource utilization) is collected from the baseline and follow-up interviews. Reported the change in number of hospitalizations per participant to week 12.
Time Frame: Baseline (LFAN Randomization), 12 weeks (LFBF)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Number analyzed (Participants) | 5 | 3 | 3
number of hospitalizations | 1.80 (1.92) | 0.67 (0.58) | 0.33 (0.58)

ADVERSE EVENTS:
Arm/Group | LFAN Placebo/LY140 mg | LFAN LY 100 mg/ LY 140 mg | LFAN LY 140 mg/LY 140 mg
Serious Adverse Events (participants affected / at risk) | 6/73 | 4/60 | 2/47
Other Adverse Events (participants affected / at risk) | 5/73 | 3/60 | 4/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LFAN Placebo/LY140 mg (N=73) | LFAN LY 100 mg/ LY 140 mg (N=60) | LFAN LY 140 mg/LY 140 mg (N=47)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Hepatic Cyst Ruptured (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LFAN Placebo/LY140 mg (N=73) | LFAN LY 100 mg/ LY 140 mg (N=60) | LFAN LY 140 mg/LY 140 mg (N=47)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Very few participants from LFBC rolled over into LFBF (N = 9). Due to insufficient sample size, the data for LFBC participants who rolled into LFBF were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days